CLINICAL TRIAL: NCT03192046
Title: Impact of Carbon Fiber AFOs on Gait and Resulting Changes in Quality of Life Across Time in Persons With PD
Brief Title: Bracing for Walking in Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: American Orthotic and Prosthetic Association (Other)
Responsible Party: Principal Investigator, Staci Shearin, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU 012014-059
Record Dates: First submitted 2017-06-13; First posted 2017-06-19 (Actual); Results first posted 2022-03-23 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-02

CONDITIONS: Gait Disorders, Neurologic; Parkinson Disease
MeSH Terms: conditions — Gait Disorders, Neurologic; Parkinson Disease

STUDY DESIGN:
Intervention Model Description: This is a randomized, repeated measures, matched group study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Carbon Fiber Ankle Foot Orthosis (AFO) (Experimental): For the bracing group, the participants will wear custom fabricated carbon fiber braces in addition to participating in a daily walking program and 7 visits of PT.
  Interventions: Device: Carbon Fiber Ankle Foot Orthosis (AFO)
- Control Group, Walking Program Only (Active Comparator): The participants in this group will be prescribed a daily home walking walking program and 7 visits of PT.
  Interventions: Other: Standardized walking/exercise program

INTERVENTIONS:
Device: Carbon Fiber Ankle Foot Orthosis (AFO) — Custom AFOs in conjunction with a walking program, working up to walking 30 minutes 6 days a week.
  Arms: Carbon Fiber Ankle Foot Orthosis (AFO)
Other: Standardized walking/exercise program — standardized walking/exercise program without any brace or AFO
  Arms: Control Group, Walking Program Only

SUMMARY:
Parkinson disease (PD) is a progressive neurological disease that results in characteristic gait dysfunction. Gait problems include decreased velocity, decreased stride length, difficulty with initiation of gait, postural stability problems and alteration in joint kinematics.1 In this typically older patient population, these gait deviations affect their participation in household and community activities. The standard of care is currently focused on therapeutic exercise and cueing of various types (visual, auditory, verbal). Current interventions have not been demonstrated to markedly improve gait kinematics, so there is a need to identify interventions that could improve gait performance in this population. Lower extremity bracing is a common and well-established intervention for gait dysfunction with other populations, including stroke and brain injury. The braces allow for improved stability, sensory feedback, and consistent tactile cues to allow patients to have the best gait mechanics with each step. It is reasonable to hypothesize that appropriate bracing may have the potential to improve gait function and kinematics in PD since these patient often have gastroc-soleus weakness. Data from our early pilot studies indicates that bracing individuals with PD can positively impact their mobility. This includes improvements in velocity, step length, and dynamic balance. Additional data supported an upward trend in quality of life.

DETAILED DESCRIPTION:
This is a randomized, repeated measures, matched group study. There will be two groups of participants, 8 participants per group, 35 participants total from time of initial enrollment in this study. Group one (G1) will receive bilateral custom braces and a standardized home walking/exercise program. Group two will receive the standardized walking/exercise program without any brace or AFO. Subjects will be randomized upon enrollment in the study. At the time of consent, random drawing from concealed envelopes with red, blue or green chips will be done to determine group assignment. Subjects will be recruited through the Clinical Center for Movement Disorders at UT Southwestern Medical Center where patients with PD receive routine evaluation and follow-up. Subjects will be followed for 6 months during this study and outcome measures will be collected 3 times over the course of the study. Subjects will be seen every 3 months for the duration of the study for testing as well as for other visits as noted in the table below. Participants will not need to have insurance benefits for initial physical therapy evaluation and for ankle braces. All subsequent visits to the Crowley gait lab for assessments and brace adjustment will be provided at no cost to the participants.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed diagnosis of Parkinson's Disease according to the UK brain bank criteria.5
2. Age between 30 and 85.
3. Measurable decrement in gait velocity (between 35 and 15 percent below age-predicted norms for self-selected walking velocity) as measured by the 6 MWT
4. Hoehn and Yahr stage 2-3.
5. Less than 10 full heel raises in single limb stance bilaterally.

Exclusion Criteria:

1. Body mass index greater than 40.
2. Passive dorsiflexion range of motion less than approximately neutral (90 degrees)
3. Any other uncontrolled health condition for which gait training is contraindicated
4. Self-report of > 1 fall/month
5. A score of 11 or less on the Short Orientation-Memory-Concentration Test of Cognitive Impairment

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Staci Shearin, Masters, Principal Investigator — UT Southwestern
Locations (1):
- UT Southwestern, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Carbon Fiber Ankle Foot Orthosis (AFO) | Control Group, Walking Program Only
Started | 5 | 4
Completed | 4 | 3
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Control Group, Walking Program Only: The participants in this group will be prescribed a daily home walking walking program and 7 visits of PT.
  Carbon Fiber Ankle Foot Orthosis (AFO): Custom AFOs in conjunction with a walking program, working up to walking 30 minutes 6 days a week.
- Total: Total of all reporting groups
Arm/Group | Carbon Fiber Ankle Foot Orthosis (AFO) | Control Group, Walking Program Only | Total
Number analyzed (Participants) | 5 | 4 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 3 | 2 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 3 | 4 | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 5 | 3 | 8
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 4 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in Gait Capacity as Assessed b 6-Minute Walk Test
Description: The 6 Minute Walk Test (6MWT) is a test of walking (gait) endurance and walking velocity and measures the distance a subject can walk indoors on a flat, hard surface in a period of 6 minutes, using assistive devices, as necessary. The test is a reliable and valid evaluation of functional exercise capacity and is used as a sub-maximal test of aerobic capacity and endurance. The test will be used to determine participant's gait efficiency at baseline and at 6 months. While the total distance covered during six minutes (6MWTD) is often used as the standard measurement of gait capacity (i.e., the maximum distance one can achieve), the endurance (i.e., ability to maintain speed over a prolonged time) can be inferred by the gait speed trajectory (GST) during the 6MW test (6MWGST).
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: Feet
Arm/Group | Carbon Fiber Ankle Foot Orthosis (AFO) | Control Group, Walking Program Only
Number analyzed (Participants) | 4 | 3
Feet | 235.7 (155.9) | 150.0 (270.0)

2. Secondary Outcome: Change in Step Length
Description: Participants will be asked to walk on a 12-16 foot long vinyl pad placed on the floor. The mat will record and analyze step length.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Carbon Fiber Ankle Foot Orthosis (AFO) | Control Group, Walking Program Only
Number analyzed (Participants) | 4 | 3
cm | 4.0 (1.8) | 0.7 (9.6)

3. Secondary Outcome: Change in Temporal Spatial Gait Parameters Using the Computerized Gait Analysis System
Description: Each subject will be asked to walk on a 12-16 foot long vinyl pad placed on the floor. The mat will record and analyze temporal and spatial gait parameters.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Deviation); unit: Cm/sec
Arm/Group | Carbon Fiber Ankle Foot Orthosis (AFO) | Control Group, Walking Program Only
Number analyzed (Participants) | 4 | 3
Cm/sec | 21.7 (18.8) | 6.26 (10.7)

ADVERSE EVENTS:
Time Frame: Adverse data was collected throughout the entire study for each participant - 6 months.
Groups:
- Carbon Fiber Ankle Foot Orthosis (AFO): For the bracing group, the participants will wear custom fabricated carbon fiber braces in addition to participating in a daily walking program and 7 visits of PT.
  Carbon Fiber Ankle Foot Orthosis (AFO): Custom AFOs in conjunction with a walking program, working up to walking 30 minutes 6 days a week.
  There were not any adverse events
- Control Group, Walking Program Only: The participants in this group will be prescribed a daily home walking walking program and 7 visits of PT.
  Carbon Fiber Ankle Foot Orthosis (AFO): Custom AFOs in conjunction with a walking program, working up to walking 30 minutes 6 days a week.
  There were not any adverse events
Arm/Group | Carbon Fiber Ankle Foot Orthosis (AFO) | Control Group, Walking Program Only
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/4
Other Adverse Events (participants affected / at risk) | 0/5 | 0/4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-02-15): https://cdn.clinicaltrials.gov/large-docs/46/NCT03192046/Prot_SAP_000.pdf